CLINICAL TRIAL: NCT05406856
Title: PROTECT: On-line Adaptive Proton Therapy for Cervical Cancer to Reduce the Impact on Morbidity and the Immune System
Brief Title: PROTECT: On-line Adaptive Proton Therapy for Cervical Cancer
Acronym: PROTECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); HollandPTC (Industry)
Responsible Party: Principal Investigator, Carien Creutzberg, prof., dr., Leiden University Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NL77911.058.21
Record Dates: First submitted 2022-05-11; First posted 2022-06-07 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Uterine Cervical Neoplasms; Locally Advanced Cervical Carcinoma
Keywords: Non-randomized phase-II trial; Primary chemoradiotherapy; Proton therapy; Organ sparing therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Cisplatin; Brachytherapy

STUDY DESIGN:
Intervention Model Description: The study is designed as a prospective, multicenter, nonrandomized phase-II-trial. During the first phase of the trial, 15 patients will be enrolled in the IMRT/VMAT treatment group. In the second phase of the trial, 15 patients will be enrolled in the IMPT group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMRT/VMAT group (Active Comparator): This group receives standard of care curative treatment with primary external beam radiation therapy (IMRT/VMAT), combined with chemotherapy, followed by 3D image (MRI)-guided adaptive brachytherapy.
  Interventions: Radiation: External beam radiation therapy: IMRT/VMAT; Drug: Cisplatin; Radiation: Brachytherapy
- IMPT group (Experimental): This group receives curative treatment with primary external beam radiation therapy (IMPT), combined with chemotherapy, followed by 3D image (MRI)-guided adaptive brachytherapy.
  Interventions: Radiation: External beam radiation therapy: IMPT; Drug: Cisplatin; Radiation: Brachytherapy

INTERVENTIONS:
Radiation: External beam radiation therapy: IMRT/VMAT — EBRT is given to a total dose of 45 Gy in 25 daily fractions of 1.8 Gy in 5 weeks. Involved nodes are boosted using a simultaneous integrated boost (SIB) to reach a total EBRT plus brachytherapy dose of 60 Gy EQD2 to provide high nodal control.
  Other Names: Intensity Modulated Radiation Therapy; Volumetric Modulated Arc Therapy
  Arms: IMRT/VMAT group
Radiation: External beam radiation therapy: IMPT — EBRT is given to a total dose of 45 Gy in 25 daily fractions of 1.8 Gy in 5 weeks. Involved nodes are boosted using a simultaneous integrated boost (SIB) to reach a total EBRT plus brachytherapy dose of 60 Gy EQD2 to provide high nodal control.
  Other Names: Intensity Modulated Proton Therapy
  Arms: IMPT group
Drug: Cisplatin — The standard chemotherapy regimen is weekly cisplatin (40 mg/m2) for 5 weeks.
Radiation: Brachytherapy — Brachytherapy is performed using a high-dose rate (HDR) after loading system to deliver a boost to any residual tumor and the cervix. Brachytherapy dose is (21-) 28 Gy in fractions of 7 Gy specified at 100% isodose around the high-risk CTV, according to the EMBRACE-II prescription protocol. The aim is to reach an equivalent dose in 2 Gy fractions including EBRT (EQD2_D90) of the high-risk CTV between 90-95 Gy, using MRI-guided adaptive brachytherapy.

SUMMARY:
This prospective, multicenter, nonrandomized phase-II-trial investigates in clinical practice the differences between intensity modulated proton therapy (IMPT) and standard intensity-modulated radiation therapy (IMRT) or volumetric-modulated arc therapy (VMAT) in the effects on dose-volume parameters and treatment-related morbidity for women with locally advanced cervical cancer undergoing chemoradiation.

DETAILED DESCRIPTION:
External beam radiation therapy (EBRT) with concurrent chemotherapy followed by brachytherapy is a highly effective treatment for locally advanced cervical cancer (LACC). However, treatment-related toxicity is common and reduces the patient's quality of life (QoL) and may affect ability to complete treatment or undergo adjuvant therapies. Intensity modulated proton therapy (IMPT) enables a significant dose reduction in organs at risk (OAR), when compared to that of standard intensity-modulated radiation therapy (IMRT) or volumetric-modulated arc therapy (VMAT). However, clinical studies evaluating whether IMPT consequently reduces side effects for LACC are lacking. The PROTECT trial is a nonrandomized prospective multicenter phase-II-trial comparing clinical outcomes after IMPT or IMRT/VMAT in LACC. Thirty women aged >18 years with a histological diagnosis of LACC will be included in either the IMPT or IMRT/VMAT group. Treatment includes EBRT (45 Gy in 25 fractions of 1.8 Gy), concurrent five weekly cisplatin (40 mg/m2), and 3D image (MRI)-guided adaptive brachytherapy. The primary endpoint is pelvic bones Dmean and mean bowel V15Gy. Secondary endpoints include dosimetric parameters, oncological outcomes, health-related QoL, immune response, safety, and tolerability. This study provides the first data on the potential of IMPT to reduce OAR dose in clinical practice and improve toxicity and QoL for patients with LACC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of cervical cancer (squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma, HPV positive or negative) with an indication for curative treatment with primary chemoradiation with concurrent cisplatin followed by 3D image-guided adaptive brachytherapy.
* Indication to include the common iliac region (minimum 5, maximum 8) or the common iliac and para-aortic regions (minimum 7, maximum 10) into the elective clinical target volume of the external beam radiotherapy.
* No distant metastasis beyond the para-aortic lymph node chain as determined by diagnostic imaging (CT or PET-CT scan)
* Age ≥ 18 years
* WHO 0-1
* Adequate systemic organ function:

  * Creatinine clearance (> 50 cc/min)
  * Adequate bone marrow function : white blood cells (WBCs) ≥3.0 x 109/l, neutrophils ≥1.5 x 109/l, platelets ≥100 x 109/l
* Patients must be accessible for treatment and follow-up
* Written informed consent according to the local Ethics Committee requirements

Exclusion Criteria:

* Small cell cancer, melanoma and other rare histological types of the cervix.
* History of another primary malignancy that could conceivably be active evaluated by the study physician. Examples of exception include, but are not limited to:

  * Malignancy treated with curative intent and with no known active disease ≥5 years.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
* Other severe diseases such as recent myocardial infarction, clinical signs of cardiac failure or clinically significant arrhythmias
* Previous pelvic or abdominal radiotherapy
* History of active primary immunodeficiency
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g. colitis or Crohn's disease])
* The use of immunosuppressive drugs at baseline
* Contraindications for weekly Cisplatin (or Carboplatin)
* Contraindications for the use of MRI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Dmean to the pelvic bones | During treatment
  Mean dose to the pelvic bones (Gy).
Mean V15Gy to the bowel | During treatment
  Mean volume of the bowel (cc) receiving 15Gy.

SECONDARY OUTCOMES:
Key dosimetric parameters of the bladder | During treatment
  Mean volume of the bladder (%) receiving greater than or equal to 15, 30, and 40Gy.
Key dosimetric parameters of the rectum | During treatment
  Mean volume of the rectum (%) receiving greater than or equal to 15, 30, and 40Gy.
Key dosimetric parameters of the sigmoid | During treatment
  Mean volume of the sigmoid (%) receiving greater than or equal to 15, 30, and 40Gy.
Key dosimetric parameters of the bowel | During treatment
  Mean volume of the bowel (cc) receiving greater than or equal to 30 and 40Gy.
Key dosimetric parameters of the body | During treatment
  Mean dose to the body (Gy) and mean volume of the body (cm3) receiving greater than or equal to 10 Gy.
Key dosimetric parameters of the pelvic bones | During treatment
  Mean volume of the pelvic bones (% or cc) receiving greater than or equal to 10, 20, and 40Gy.
Key dosimetric parameter of the kidneys | During treatment
  Mean dose to the kidneys (Gy).
Key dosimetric parameters of the spinal cord | During treatment
  Mean volume of the spinal cord (%) receiving greater than or equal to 15 and 30Gy.
Other dosimetric parameters of critical organs | During treatment
  Mean volume of an organ at risk (% or cc) receiving greater than or equal to xGy.
Overall survival | At Month 12 after end of treatment
  The percentage (%) of included patients who are alive after start of treatment
Complete response | At Month 3 after end of treatment
  Absence of disease in the cervix, uterus, upper vagina, and parametria.
Pelvic recurrence-free survival | At Month 12 after end of treatment
  The time from start of treatment to the first occurrence of pelvic recurrence.
Distant recurrence-free survival | At Month 12 after end of treatment
  The time from start of treatment to the first occurrence of distant recurrence.
Health-related Quality of Life | At baseline, week 4 of EBRT, end of treatment, and at Month 3, Month 6, Month 9, and Month 12 after end of treatment
  For the evaluation of patient reported symptoms and QoL, the European Organization for Research and Treatment of Cancer (EORTC)-core (C-30) questionnaire, the CX24 module for cervical cancer, and six additional questions from EN24 module will be used.
Safety and tolerability (toxicity) | At baseline, week 4 of EBRT, end of treatment, and at Month 3, Month 6, Month 9, and Month 12 after end of treatment
  Toxicity will be graded according to the NCI-CTCAE version 5.0.
The effect on the local immune system (analyzed with the Nanostring PanCancer IO 360 panel) | At baseline and at the first brachytherapy session
  Tumor biopsies will be collected for evaluation of the impact of treatment on the local immune response.
The effect on the systemic immune system | At baseline, week 4 of treatment, and at Month 1, Month 2, Month 3, and Month 12 after end of treatment
  Blood samples will be collected for immune-monitoring. Full blood count, peripheral blood mononuclear cells, leukocyte differentiation, APC quality, T cell reactivity, and immune composition changes will be measured.
The effect on bone marrow fat fraction | At baseline, for brachytherapy purposes, and at Month 3 and Month 12 after end of treatment.
  Patients will have an MR scan with Dixon technique for evaluation of bone marrow fat fraction in the vertebral column and femoral necks.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie M. de Boer, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
After completion of the trial and publication of the final results, data will be available upon request with a scientific proposal. Approval by the trial management group is necessary.
Supporting Information: Study Protocol, CSR
Time Frame: After final publication
Access Criteria: Approval by the trial management group is necessary

REFERENCES:
- [Background] Corbeau A, Nout RA, Mens JWM, Horeweg N, Godart J, Kerkhof EM, Kuipers SC, van Poelgeest MIE, Kroep JR, Boere IA, van Doorn HC, Hoogeman MS, van der Heide UA, Putter H, Welters MJP, van der Burg SH, Creutzberg CL, de Boer SM. PROTECT: Prospective Phase-II-Trial Evaluating Adaptive Proton Therapy for Cervical Cancer to Reduce the Impact on Morbidity and the Immune System. Cancers (Basel). 2021 Oct 15;13(20):5179. doi: 10.3390/cancers13205179. PMID 34680328